CLINICAL TRIAL: NCT03050320
Title: Improving Resilience and Longevity for Workers Through Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Workplace Exercise
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Resilience; Exercise in the workplace
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The participants in this arm will be asked to attend 3 group classes per week for 12 weeks taught by a certified exercise instructor. Five class times will be offered per week. These classes included a warm-up, static poses shown to decrease knee joint loading, and a cool down including flexibility exercises. Measurements will be obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes included clinical mobility; pain; isometric leg strength; cardiovascular fitness; and resilience.
  Interventions: Other: Exercise
- No Exercise (Other): The participants in this arm will be asked to refrain from changing their physical activity over the 12 weeks and maintain any strategies typically used to manage knee and/or hip pain. Since it is known that exercise is beneficial for pain management and strengthening in knee OA, participants randomized to the no exercise group will be offered the same exercise program following completion of the study. Measurements will be obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes included clinical mobility; pain; isometric leg strength; cardiovascular fitness; and resilience.
  Interventions: Other: No Exercise

INTERVENTIONS:
Other: Exercise — A biomechanical exercise program shown to decrease joint loading will be administered 3 times a week for 12 weeks. Outcomes included mobility performance; pain; strength; cardiovascular fitness; and resilience.
  Arms: Exercise
Other: No Exercise — A no exercise (control) group will be asked to maintain their existing activity level for 12 weeks. Outcomes included mobility performance; pain; strength; cardiovascular fitness; and resilience.
  Arms: No Exercise

SUMMARY:
The purpose of this study is to examine the impact of an OA-specific aerobic and strengthening exercise program, delivered within the workplace, on mobility, pain, physical capacity, and resilience among workers with knee or hip OA as well as those with no joint pain. The investigators hypothesize that exercise designed for OA, delivered at work, will improve all of these outcomes.

DETAILED DESCRIPTION:
The Canadian workforce is aging. The most prevalent age group is 50-54 years and most of these Canadians will aim to continue working over the next 10 years. However, the impact of arthritis on aging Canadians compromises their ability to continue working. By 2031, over 2 million Canadians aged 45 to 64 years will have arthritis. The investigators aim to boost the ability of adults with the most common arthritis, osteoarthritis (OA), as well as adults without OA, to engage in the workforce for as long as they desire. Identifying strategies to promote productivity among workers with knee and hip OA will be of great public health significance in the coming decades. However, the investigators face two challenges. First, obesity among sedentary workers is a risk for worsening knee and hip OA. Second, large occupational loads on the knee and hip worsen OA. Exercise has the most promise in addressing these challenges because it reduces pain and sick time, and improves mental health. Thus, there is a call for studies examining exercise for workers with knee and hip OA.

ELIGIBILITY:
Inclusion Criteria:

* full-time or part-time administrative employees

Exclusion Criteria:

* Any other forms of arthritis
* Osteoporosis-related fracture
* History of patellofemoral symptoms
* Active non-arthritic hip or knee disease
* Hip or knee surgery
* Use of cane or walking aid
* Unstable heart condition
* Neurological conditions
* Hip, knee or ankle injuries in past 3 months
* Physician-advised restriction to physical activity
* Any injuries that would prohibit participation in exercise
* Ipsilateral ankle conditions
* Currently receiving cancer treatment
* Currently pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Maly, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulla DM, Wiebenga EG, Chopp-Hurley JN, Kaip L, Jarvis RS, Stephens A, Keir PJ, Maly MR. The Effects of Lower Extremity Strengthening Delivered in the Workplace on Physical Function and Work-Related Outcomes Among Desk-Based Workers: A Randomized Controlled Trial. J Occup Environ Med. 2018 Nov;60(11):1005-1014. doi: 10.1097/JOM.0000000000001408. PMID 30020219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | No Exercise
Started | 21 | 22
Completed | 20 | 21
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: There were no cross overs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | No Exercise | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.5) | 43.3 (10.4) | 43.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 21 | 22 | 43
Type of Osteoarthritis [Count of Participants; unit: Participants]
  Hip Osteoarthritis | 1 | 0 | 1
  Knee Osteoarthritis | 2 | 3 | 5
  No Osteoarthritis | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Functional Scale
Description: The Lower Extremity Function Scale (LEFS) consists of 20 items, on an adjectival scale, that assess difficulty during mobility tasks ranging from transfers to running. Each item is scored from 0 (extreme difficulty or unable to perform activity), to 4 (no difficulty to perform activity). The minimum possible score is 0, and the maximum possible score is 80. Scores closer to 80 represent better self-reported physical function. It is reliable and valid in knee OA and has superior sensitivity to change compared to similar measures
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale | 5.3 (9.0) | -1.6 (8.5)

2. Secondary Outcome: Change in Self-reported Knee and Hip Pain
Description: Change in self-reported knee and hip pain will be assessed with 3 valid and reliable questionnaires: the Knee injury and Osteoarthritis Outcome Score (KOOS), the Hip disability and Osteoarthritis Outcome Score (HOOS), and the Intermittent and Constant Osteoarthritis Pain (ICOAP) score. The KOOS and HOOS pain scores represent a normalized score from 0 (extreme symptoms) to 100 (no symptoms). KOOS and HOOS scores closer to 100 indicate fewer symptoms. The ICOAP consists of two sub-scales: constant pain (5 items) and intermittent pain (6 items). The score from each subscale represents a normalized score from 0 (no pain) to 100 (extreme pain). ICOAP scores closer to 0 indicate less pain. The items from each subscale are averaged to produce a normalized ICOAP total score, ranging from 0 (no pain) to 100 (extreme pain).
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale
  KOOS Pain | 3.3 (7.2) | -0.1 (3.8)
  HOOS Pain | 5.4 (12.3) | 2.1 (6.7)
  ICOAP Constant Pain | -0.8 (10.0) | 0.2 (4.0)
  ICOAP Intermittent Pain | -6.1 (15.5) | -2.4 (9.0)
  ICOAP Total | -3.6 (11.4) | -1.2 (5.9)

3. Secondary Outcome: Change in Self-reported Upper Extremity Pain
Description: The Disabilities of the Arm Shoulder and Hand is a 30-item questionnaire addressing upper extremity physical function and symptoms. The DASH is suitable for people with any upper limb musculoskeletal disorders and can also monitor changes in severity of symptoms and functional abilities over time. Each item is scored from 1 (no difficulty) to 5 (unable). Total scores range from 0 to 100, with higher scores indicating more upper limb problems.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale | -1.6 (5.4) | 0.2 (4.1)

4. Secondary Outcome: Change in Isometric Knee Extensor and Flexor Strength
Description: The peak torque developed during knee extension and flexion during a maximum isometric contraction will be measured by use of a ergoFET hand-held dynamometer.
Time Frame: Weeks 1 and 13
Population: Data from one individual from the No Exercise group was not collected for this measure due to an unrelated back injury.
Measure: Mean (Standard Deviation); unit: Newton*meters/kg
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 20
Newton*meters/kg
  Extension | 0.15 (0.29) | 0.00 (0.28)
  Flexion | 0.07 (0.11) | 0.00 (0.14)

5. Secondary Outcome: Change in Grip Strength
Description: Grip strength will be assessed using a Jamar hand dynamometer. The hand dynamometer will be set to a fixed position and all values of grip force will be expressed in kg.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Kg of force
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Kg of force
  Dominant hand | -0.4 (5.5) | 0.9 (5.1)
  Non-dominant hand | -0.9 (4.9) | 1.6 (3.4)

6. Secondary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness will be calculated using the Single Stage Treadmill Walking Test. Predictions of VO2max will be made from heart rate (measured with a heart rate monitor), walking speed, age and gender.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
mL/kg/min | 1.0 (1.9) | 0.1 (1.8)

7. Secondary Outcome: Change in Mobility Performance (Six-Minute Walk Test)
Description: Mobility performance will be measured using the Six-Minute Walk Test (6MWT). For this test, participants are instructed to walk as far as possible in 6 minutes. The distance covered in 6 minutes is recorded in metres. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Weeks 1 and 13
Population: Data from one individual from the No Exercise group was not collected for this measure due to an unrelated back injury.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 20
Meters | 36.8 (51.6) | 18.4 (29.6)

8. Secondary Outcome: Change in Mobility Performance (Stair Ascent and Descent)
Description: Mobility performance will be measured using the Stair Ascent and Descent Test. For this test, the time taken to ascend, as well as descend nine stairs is recorded in seconds. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Weeks 1 and 13
Population: Data from one individual from the No Exercise group was not collected for this measure due to an unrelated back injury.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 20
Seconds
  Stair Ascent | -0.5 (0.8) | -0.1 (0.5)
  Stair Descent | -0.6 (1.1) | 0.0 (0.5)

9. Secondary Outcome: Change in Mobility Performance (30-second Chair Stand Test)
Description: Mobility performance will be measured using the 30-second Chair Stand Test. This test measures the number of times participants can rise and lower from a standard height chair, without using arm rests, in a 30-second period.This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Weeks 1 and 13
Population: Data from one individual from the No Exercise group was not collected for this measure due to an unrelated back injury.
Measure: Mean (Standard Deviation); unit: Number of chair stands
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 20
Number of chair stands | 3.5 (3.2) | 1.6 (2.9)

10. Secondary Outcome: Change in Resilience
Description: Resilience will be measured using the Resilience Scale 25 Survey, which is a 25-item questionnaire designed to evaluate a participants ability to adapt to stress and adversity. The test is scored out of 175 (scores ranging from 25 to 175), with higher scores indicating higher resilience.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale | 8.6 (10.5) | 3.3 (9.6)

11. Secondary Outcome: Change in Work Ability
Description: The Work Ability Index (WAI) is a widely-used self-report questionnaire that evaluates a worker's capacity to perform a job accounting for their physical and mental well-being in addition to the demands of their job. The WAI consists of seven dimensions including current work ability relative to life-time best, work ability related to job demands, number of current physician-diagnosed health conditions, estimated work impairment due to the conditions, sick leave over the past year, own prognosis, and mental resources. Total scores range from 7 to 49 and can fall under one of four classifications: poor work ability that should be restored (7-27), moderate work ability that should be improved (28-36), good work ability that should be supported (37-43), and excellent work ability that should be maintained (44-49). The WAI produces reliable data.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale | 0.9 (3.3) | 0.6 (2.9)

12. Secondary Outcome: Change in Depressive Symptoms
Description: Depression will be assessed with the Centre of Epidemiological Studies Depression (CES-D) Scale, a 20-item scale developed for the general population with emphasis on affect. Elements of affect include mood, guilt, worthlessness, helplessness, appetite, and sleep. Each item is scored from 0 (rarely or none of the time), to 3 (most of the time). The items are summed to produce a total score between 0 and 60 with a score of 16 or higher indicating depression.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale | 1.0 (4.8) | -0.1 (4.5)

13. Secondary Outcome: Change in Arthritis-related Self-Efficacy
Description: The Arthritis Self-Efficacy Scale (ASES) measures arthritis-specific beliefs regarding perception of performance on certain tasks to cope with the disease. The ASES is measured using 20 questions on a 10-100 scale with respect to three main areas: pain management (5 questions), physical function (9 questions), and other symptoms (6 questions). Each question is scored from 10 (very uncertain), to 100 (very certain), in 10-point increments. The minimum score for each subscale is 10, and the maximum score for each subscale is 100. The scores from each subscale are averaged to produce a normalized total score. Scores closer to 100 indicate greater certainty that a participant can cope with a particular task as a consequence of their disease.
Time Frame: Weeks 1 and 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 20 | 21
Units on a scale
  Pain | 0.1 (1.6) | -0.4 (2.0)
  Function | 0.2 (0.5) | 0.1 (0.5)
  Symptom | 0.5 (1.7) | 0.1 (1.7)
  Total | 0.8 (3.3) | -0.2 (3.0)

ADVERSE EVENTS:
Time Frame: Week 1 and week 13.
Arm/Group | Exercise | No Exercise
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

LIMITATIONS AND CAVEATS:
* a limited number of participants were recruited due to time and space limitations within the exercise facility
* physical activity levels of the control group during the 12-week intervention period were not quantified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03050320/Prot_SAP_ICF_000.pdf